CLINICAL TRIAL: NCT07337356
Title: Research on the Development and Validation of an Early Prediction Model for Delirium Based on Machine Vision Analysis
Brief Title: Research on the Development and Validation of an Early Prediction Model for Delirium
Status: Not yet recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZWQ21886-2025-EC-579
Record Dates: First submitted 2026-01-04; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Delirium; Prediction Models; Machine Learning
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- observational: 1. Meets the delirium diagnostic criteria specified in the Diagnostic and Statistical Manual of Mental Disorders (5th Edition) (DSM-5), which requires the concurrent presence of: ① disturbance in awareness (reduced clarity of awareness of the environment) ; ② change in cognition (e.g., memory impairment, disorientation);
  2. Undergoes consecutive daily assessments for 7 days using the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) at three time points (8:00, 14:00, 20:00) with an interval of ≥ 6 hours between each assessment, with at least two positive results;
- control: Admitted to the ICU during the same period, with negative results on consecutive daily CAM-ICU assessments for 3 days (three assessments per day as the observational group).

SUMMARY:
Delirium has a high incidence rate and significantly affects patient prognosis. Diagnosis often relies on manual assessment, which is subject to strong subjectivity, high rates of missed diagnosis, and poor stability. This study employs non-contact identification technology based on machine vision analysis to quantitatively analyze characteristic biological feature data such as micro-expressions. It then investigates the correlation between these features and delirium subtypes. By integrating clinical phenotypic data and using machine learning algorithms, a multi-modal early prediction model for delirium is constructed to meet the clinical need for early warning of delirium subtypes and enhance the efficacy of delirium identification.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, expected ICU stay ≥ 24 hours, and informed consent to participate in this study;

Exclusion Criteria:

* Patients with severe facial trauma/deformities that prevent complete expression acquisition, and patients with a history of emotional problems (such as anxiety, depression, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years old) admitted to the ICU of Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, including elderly patients, those post-surgery, with sepsis, and trauma, which are common high-risk populations for delirium.
Sampling Method: Non-Probability Sample
Enrollment: 795 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with delirium as assessed by DSM-5 | 7th day after ICU admission
  Zero is equivalent to no delirium and a high score means a higher occurrence of delirium

SECONDARY OUTCOMES:
Accuracy | 7th day after ICU admission
  Zero is equivalent to the minimum accuracy, while a value of 1 represents perfect accuracy
Precision | 7th day after ICU admission
  The proportion of truly positive samples among those predicted as positive; the closer the score is to 1, the higher the precision
Recall | 7th day after ICU admission
  The proportion of truly positive samples that are correctly predicted; the closer the score is to 1, the higher the diagnostic sensitivity
F1-score | 7th day after ICU admission
  The harmonic mean of precision and recall; the higher the score, the better the diagnostic performance of the model

IPD SHARING:
Plan to Share IPD: No